CLINICAL TRIAL: NCT06168422
Title: A Cohort Study of PCI Strategies for Severely Calcified Lesions of Complex Coronary Arteries in the Elderly
Acronym: PSSCCE
Status: Recruiting | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Other Study IDs: HenanICE202312
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DES Group: All lesions in these patients were treated with DES
  Interventions: Device: DES
- DES+DCB Group: These patients were treated using a combination of DES and DCB
  Interventions: Device: DES; Device: DCB
- DCB Group: All lesions in these patients were treated with DCB
  Interventions: Device: DCB

INTERVENTIONS:
Device: DES — drug eluting stent
  Groups: DES Group; DES+DCB Group
Device: DCB — drug-coated balloon
  Groups: DCB Group; DES+DCB Group

SUMMARY:
The aim of this observational study is to compare the prognostic outcomes of various PCI strategies in elderly patients with complex coronary calcified lesions. The patients will be classified into two groups and assigned different PCI strategies, either stenting or stenting combined with pharmacologic balloon implantation. The investigators will assess the one-year prognosis for major adverse cardiovascular events in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years;
2. Meet the indications for coronary intervention;
3. IVUS examination suggests severe calcified lesions (calcification angle >270°) or OCT examination suggests severe calcified lesions (calcification angle >180° and/or length >5mm and/or thickness >0.5mm);
4. The diameter of the target lesion vessel is greater than 2.75mm;
5. The total length of the lesion is more than 60mm and/or the number of lesions to be treated is ≥3 and/or the number of vessels to be treated is ≥2.

Exclusion Criteria:

1. inability to provide written informed consent;
2. inability to administer antiplatelet agents and anticoagulant therapy;
3. the subject is participating in other unfinished clinical trials;
4. life expectancy <1 year;
5. non-in situ vascular lesions;
6. patients with haemodynamic instability;
7. Previous stroke within 6 months.
8. left main stem lesions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients with calcified coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
MACEs | 12 months
  A Composite Event Including Cardiac Death, Myocardial Infarction, Stroke, and Target Vessel Revascularization

SECONDARY OUTCOMES:
Cardiac Death | 12 months
  Cardiac Death
Myocardial Infarction | 12 months
  Myocardial Infarction
Target Vessel Revascularization | 12 months
  Target Vessel Revascularization
Stroke | 12 months
  Stroke
BRCA 2,3-5 | 12 months
  BRCA 2,3-5

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, Principal Investigator — Fuwai central China cardiovascular hospotial
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided